CLINICAL TRIAL: NCT01436643
Title: A 21-week, Multicenter, Open Label Study to Evaluate the Safety and Tolerability Profile of the Combination of a SSRI or SNRI Antidepressive Therapy With Oral Fingolimod in the Treatment of RRMS Patients With Mild to Moderate Depression
Brief Title: Combination of Antidepressants and Fingolimod Relapsing-remitting Multiple Sclerosis (RRMS) Patients With Depression
Acronym: REGAIN
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to slow enrollment the study was terminated early
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CFTY720DDE06; 2011-001692-39 (EudraCT Number)
Record Dates: First submitted 2011-09-16; First posted 2011-09-20 (Estimated); Results first posted 2014-09-25 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Depression; Relapsing-remitting Multiple Sclerosis
Keywords: Depression; Multiple Sclerosis; Fingolimod; Venlafaxine; Fluoxetine
MeSH Terms: conditions — Depression; Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — Venlafaxine Hydrochloride; Fluoxetine; Citalopram; Fingolimod Hydrochloride

ARMS (3):
- Fluoxetine and Fingolimod (Experimental): Fingolimod 0.5 mg per capsule(hard gelatin capsules) was taken p.o. once daily. Fluoxetine, supplied in blistered packs containing 20 tablets; starting dose 20 mg; final dose 40 mg
  Interventions: Drug: Fluoxetine; Drug: Fingolimod
- Venlafaxine and Fingolimod (Experimental): Fingolimod 0.5 mg per capsule(hard gelatin capsules) was taken p.o. once daily. Venlafaxine, supplied in blistered packs containing 14 capsules; starting dose 75 mg; final dose 150 mg
  Interventions: Drug: Venlafaxine; Drug: Fingolimod
- Citalopram and Fingolimod (Experimental): Fingolimod 0.5 mg per capsule(hard gelatin capsules) was taken p.o. once daily. Citalopram, supplied in blistered packs containing 20 tablets; starting dose 20 mg, final dose 40 mg
  Interventions: Drug: Citalopram; Drug: Fingolimod

INTERVENTIONS:
Drug: Venlafaxine — Venlafaxine starting dose was 75 mg and given once daily for at least 7 days and a maximum of 28 days. Dosage was increased afterwards to the individual final dose given once daily, i.e. after at least 7 days and a maximum of 28 days, patients were titrated to their maximum dose of 150 Mg
  Arms: Venlafaxine and Fingolimod
Drug: Fluoxetine — Fluoxetine starting dose was 20 mg and given once daily for at least 7 days and a maximum of 28 days. Dosage was increased afterwards to the individual final dose given once daily, i.e. after at least 7 days and a maximum of 28 days, patients were titrated to their maximum dose of 40 Mg
  Arms: Fluoxetine and Fingolimod
Drug: Citalopram — Citalopram starting dose was 20 mg and given once daily for at least 7 days and a maximum of 28 days. Dosage was increased afterwards to the individual final dose given once daily, i.e. after at least 7 days and a maximum of 28 days, patients were titrated to their maximum dose of 40 Mg
  Arms: Citalopram and Fingolimod
Drug: Fingolimod — Dosage of 0.5 mg per capsule (hard gelatin capsules) was taken p.o. once daily. Fingolimod was supplied in bottles containing 35 capsules each.

SUMMARY:
This is a prospective, multi-center, open-label study in Relapsing-remitting Multiple Sclerosis (RRMS) patients with mild to moderate depression treated with selected serotonin reuptake inhibitors (SSRI) or serotonin and norepinephrine reuptake inhibitors (SNRI) antidepressants over 16 weeks as add-on to fingolimod treatment. It is designed to evaluate the safety and tolerability of this combination in this patient population based on an immunomodulatory treatment with fingolimod.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with relapsing remitting MS defined by 2010 revised McDonald criteria (see Appendix 4)
* Patients with Expanded Disability Status Scale (EDSS) score of 0-6.5 (see Appendix 8)
* Patients with high disease activity despite treatment with a disease modifying therapy (> 1 relapse in the previous year, > 9 hyperintense T2 lesions or > 1 Gd-enhancing lesion or "non-responding" which could be defined as unchanged or increased relapse rate or ongoing severe relapses compared to previous year)or patients with rapidly evolving severe RRMS (e.g. > 2 relapses with disease progression in one year and > 1 Gd-enhancing lesion or with a significant increase in T2 lesions compared to a recent MRI)
* Depression according to ICD-10 criteria
* Mild-moderate depression assessed by BDI-II score between 14-28 inclusively measured before study inclusion and before fingolimod is administered

Exclusion Criteria:

* Patients with a history of chronic disease of the immune system other than MS which requires systemic immunosuppressive treatment, or a known immunodeficiency syndrome. Patients with Crohns disease or ulcerative colitis are excluded without exception
* History or presence of malignancy (other than localized basal or squamous cell carcinoma of the skin)
* Patients with active systemic bacterial, viral or fungal infections, or known to have AIDS, Hepatitis B, Hepatitis C infection or to have positive HIV antibody, Hepatitis B surface antigen or Hepatitis C antibody tests
* Negative for varicella-zoster virus IgG antibodies at Screening
* Patients who expect to be treated with any disease modifying drugs (DMD) during the study (i.e. IFN-β, glatiramer acetate); however no washout is needed for DMDs prior to start of fingolimod
* Patients who are or have been treated with:
* immunoglobulins and/or monoclonal antibodies (including natalizumab) within 3 months prior to start of fingolimod
* Systemically applied corticosteroids or adrenocorticotropic hormones (ACTH) within 1 month prior to start of fingolimod (nevertheless, topical application is permitted);
* Immunosuppressive medications such as azathioprine or methotrexate, within 3 months prior to start of fingolimod;
* Cyclophosphamid and mitoxantrone within 6 months prior to start of fingolimod
* cladribine at any time
* current psychological or pharmacological treatment for depression (MAO inhibitors in particular), a washout period of 1 month prior start of fingolimod is required
* current treatment with linezolid, a washout period of 1 month prior start of fingolimod is required

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2011-11; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (24):
- Germany (24):
  - Novartis Investigative Site, Altenholz-Stift, Germany
  - Novartis Investigative Site, Achim
  - Novartis Investigative Site, Aschaffenburg
  - Novartis Investigative Site, Bad Honnef
  - Novartis Investigative Site, Baesweiler
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bielefeld
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Bremerhaven
  - Novartis Investigative Site, Butzbach
  - Novartis Investigative Site, Grevenbroich
  - Novartis Investigative Site, Heidenheim
  - Novartis Investigative Site, Klingenmünster
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Merzig
  - Novartis Investigative Site, Nienburg
  - Novartis Investigative Site, Oberhausen
  - Novartis Investigative Site, Oldenburg
  - Novartis Investigative Site, Potsdam
  - Novartis Investigative Site, Schwalmstadt-Treysa
  - Novartis Investigative Site, Stadtroda
  - Novartis Investigative Site, Tübingen
  - Novartis Investigative Site, Weil am Rhein
  - Novartis Investigative Site, Zwickau

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The safety set was used for analysis, which consists of 54 patients, of whom 2 patients did not start treatment with any antidepressant
Groups:
- Pre-treatment With Fingolimod: During 2weeks pre-treatment period patients received Fingolimod 0.5 mg per capsule (hard gelatin capsules) orally once daily.
Period: 2-week Pre-treatment
Arm/Group | Fluoxetine and Fingolimod | Venlafaxine and Fingolimod | Citalopram and Fingolimod | Pre-treatment With Fingolimod
Started | 0 | 0 | 0 | 54
Completed | 0 | 0 | 0 | 44
Not Completed | 0 | 0 | 0 | 10
Not completed — Abnormal test result | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 5
Not completed — Protocol Violation | 0 | 0 | 0 | 4
Period: Core Phase (16 Weeks)
Arm/Group | Fluoxetine and Fingolimod | Venlafaxine and Fingolimod | Citalopram and Fingolimod | Pre-treatment With Fingolimod
Started | 17 | 15 | 20 | 0
Completed | 16 | 11 | 17 | 0
Not Completed | 1 | 4 | 3 | 0
Not completed — Adverse Event | 0 | 3 | 1 | 0
Not completed — Abnormal Test result | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 1 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The safety set was used for analysis, which consists of 54 patients, of whom 2 patients did not start treatment with any antidepressant
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluoxetine and Fingolimod | Venlafaxine and Fingolimod | Citalopram and Fingolimod | Total
Number analyzed (Participants) | 17 | 15 | 20 | 52
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.2 (9.22) | 40.0 (9.28) | 41.2 (10.22) | 41.8 (9.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 10 | 17 | 42
  Male | 2 | 5 | 3 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Adverse Events, Serious Adverse Events and Death
Description: In this analysis patients with all (serious and non-serious) adverse events, and death were reported.
  See Safety Section.
Time Frame: 21 weeks
Population: as for baseline characteristics
Measure: Number; unit: Participants
Groups:
- Fingolimod: 2 Week Pre-treatment Period: Fingolimod 0.5 mg per capsule (hard gelatin capsules) was taken p.o. once during 2 week pre-treatment period.
Arm/Group | Fluoxetine and Fingolimod | Venlafaxine and Fingolimod | Citalopram and Fingolimod | Fingolimod
Number analyzed (Participants) | 17 | 15 | 20 | 54
Participants
  Any Adverse Event | 11 | 12 | 12 | 15
  Death | 0 | 0 | 0 | 0
  Serious Adverse Event | 0 | 1 | 1 | 1

ADVERSE EVENTS:
Description: The safety set (SS) consists of all enrolled patients for whom safety information was collected. Of note, the statement that a patient had no adverse events also constitutes a safety assessment. Fingolimod 2 week pretreatment included 2 patients who did not receive antidepressant.
Arm/Group | Fingolimod | Venlafaxine and Fingolimod | Citalopram and Fingolimod | Fluoxetine and Fingolimod
Serious Adverse Events (participants affected / at risk) | 1/54 | 1/15 | 1/20 | 0/17
Other Adverse Events (participants affected / at risk) | 15/54 | 12/15 | 12/20 | 11/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fingolimod (N=54) | Venlafaxine and Fingolimod (N=15) | Citalopram and Fingolimod (N=20) | Fluoxetine and Fingolimod (N=17)
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 1 | 0 | 0 | 0
MULTIPLE SCLEROSIS RELAPSE (Nervous system disorders) | 0 | 1 | 0 | 0
SUICIDAL IDEATION (Psychiatric disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fingolimod (N=54) | Venlafaxine and Fingolimod (N=15) | Citalopram and Fingolimod (N=20) | Fluoxetine and Fingolimod (N=17)
LYMPHOPENIA (Blood and lymphatic system disorders) | 6 | 0 | 0 | 0
TACHYCARDIA (Cardiac disorders) | 0 | 1 | 0 | 0
ASTHENOPIA (Eye disorders) | 0 | 0 | 0 | 1
CONJUNCTIVAL HAEMORRHAGE (Eye disorders) | 0 | 0 | 0 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 0 | 0 | 1
CONSTIPATION (Gastrointestinal disorders) | 0 | 1 | 1 | 0
DIARRHOEA (Gastrointestinal disorders) | 0 | 1 | 1 | 0
DRY MOUTH (Gastrointestinal disorders) | 0 | 0 | 0 | 1
GASTROINTESTINAL DISORDER (Gastrointestinal disorders) | 0 | 0 | 0 | 1
NAUSEA (Gastrointestinal disorders) | 0 | 3 | 4 | 4
TOOTHACHE (Gastrointestinal disorders) | 0 | 1 | 0 | 0
FATIGUE (General disorders) | 0 | 1 | 0 | 2
FEELING HOT (General disorders) | 0 | 1 | 0 | 0
OEDEMA PERIPHERAL (General disorders) | 0 | 0 | 1 | 0
PAIN (General disorders) | 0 | 0 | 0 | 1
THIRST (General disorders) | 0 | 0 | 0 | 1
BRONCHITIS (Infections and infestations) | 0 | 0 | 1 | 1
GASTROINTESTINAL INFECTION (Infections and infestations) | 0 | 0 | 0 | 1
INFLUENZA (Infections and infestations) | 0 | 1 | 0 | 1
NASOPHARYNGITIS (Infections and infestations) | 2 | 1 | 1 | 2
RHINITIS (Infections and infestations) | 0 | 0 | 1 | 0
TONSILLITIS (Infections and infestations) | 0 | 1 | 0 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 0 | 1 | 0
CONTUSION (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
FALL (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
BLOOD BILIRUBIN INCREASED (Investigations) | 0 | 0 | 0 | 1
ELECTROCARDIOGRAM ABNORMAL (Investigations) | 1 | 0 | 1 | 0
LABORATORY TEST ABNORMAL (Investigations) | 1 | 1 | 1 | 1
WEIGHT DECREASED (Investigations) | 0 | 1 | 0 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
SKIN PAPILLOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
DIZZINESS (Nervous system disorders) | 0 | 1 | 1 | 0
DYSGEUSIA (Nervous system disorders) | 0 | 1 | 0 | 0
HEADACHE (Nervous system disorders) | 1 | 1 | 1 | 2
HYPOAESTHESIA (Nervous system disorders) | 0 | 1 | 0 | 0
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 0 | 1 | 0 | 0
MULTIPLE SCLEROSIS RELAPSE (Nervous system disorders) | 2 | 2 | 0 | 2
OPTIC NEURITIS (Nervous system disorders) | 0 | 0 | 0 | 1
PAROSMIA (Nervous system disorders) | 0 | 1 | 0 | 0
SEDATION (Nervous system disorders) | 0 | 0 | 1 | 0
SOMNOLENCE (Nervous system disorders) | 1 | 1 | 0 | 0
TREMOR (Nervous system disorders) | 0 | 0 | 0 | 1
AGITATION (Psychiatric disorders) | 0 | 0 | 0 | 1
INSOMNIA (Psychiatric disorders) | 1 | 2 | 0 | 0
LIBIDO DISORDER (Psychiatric disorders) | 0 | 1 | 0 | 0
SLEEP DISORDER (Psychiatric disorders) | 0 | 0 | 1 | 0
EJACULATION DISORDER (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
METRORRHAGIA (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
YAWNING (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
ALOPECIA (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
DERMATITIS ALLERGIC (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 1
SKIN LESION (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
FLUSHING (Vascular disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.